CLINICAL TRIAL: NCT04958122
Title: Clinical Trial Comparing the Effectiveness of Cefixime Versus Penicillin G for Treatment of Early Syphilis
Brief Title: Cefixime Clinical Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: AIDS Healthcare Foundation (Other); Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Jeffrey D Klausner, Clinical Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-21-00288
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Syphilis; Human Immunodeficiency Virus
Keywords: Cefixime; Treponema pallidum; Penicillin; Early Syphilis
MeSH Terms: conditions — Syphilis; Acquired Immunodeficiency Syndrome; Treponemal Infections | interventions — Cefixime; Penicillin G Benzathine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cefixime (Experimental): Oral cefixime 400mg, taken twice a day for 10 days
  Interventions: Drug: Cefixime 400mg
- Benzathine Penicillin G (Active Comparator): Single intramuscular injection of 2.4 million units of benzathine penicillin G
  Interventions: Drug: benzathine penicillin

INTERVENTIONS:
Drug: Cefixime 400mg — Oral cefixime 400 mg, one capsule, twice a day for 10 days
  Other Names: supprax
  Arms: Cefixime
Drug: benzathine penicillin — Standard of care benzathine penicillin G, one intramuscular injection, 2.4MU
  Other Names: bicillin
  Arms: Benzathine Penicillin G

SUMMARY:
This study aims to evaluate the efficacy of cefixime compared to benzathine penicillin G in the treatment of syphilis.

DETAILED DESCRIPTION:
This will be a randomized, multisite, open-label, non-inferiority clinical trial to evaluate the effectiveness of cefixime (400mg orally, twice a day, for 10 days) compared to benzathine penicillin G (2.4 million units, intramuscularly) in patients with and without HIV infection. In total, 400 participants with early syphilis will be enrolled from 9 clinical sites in the U.S. and Peru. Participants will participate in follow-ups to monitor clinical outcomes and serological response (RPR titer) every 3 months for 9 months. Study findings may identify an efficacious alternative syphilis treatment to penicillin, effective for people living with HIV infection, to help address the crisis of penicillin shortages and offer options for those with penicillin allergy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of primary, secondary, or early latent syphilis with RPR titer ≥1:8 within 3 weeks prior to enrollment
* 18 years of age or older
* Able to provide informed consent
* Individuals with HIV infection must be on treatment for HIV infection and virologically suppressed (viral load <200 copies/mL) or have a CD4 count ≥ 350 cells/mm3 according to most recent labs before study enrollment

Exclusion Criteria:

* Pregnancy or a positive pregnancy test on the day of enrollment
* Patients showing signs and symptoms of neurosyphilis
* Serofast RPR titer, defined as persistently positive RPR titer without more than 4-fold (2-titer level) change for 12 months or greater
* Recent (within the past 7 days) or concomitant antimicrobial therapy with activity against syphilis, namely azithromycin, doxycycline, ceftriaxone, or other beta-lactam antibiotics (e.g. amoxicillin)
* Individuals with HIV infection who report HIV treatment interruption for more than 4 weeks since their most recent viral load or CD4 test
* Self-reported allergy to cephalosporins or penicillin
* Unwilling or unable to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Response to treatment | 6 months
  Percentage of cefixime participants with a 4-fold decrease or greater in the serum RPR titer 3 or 6 months after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Klausner, MD MPH, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers